CLINICAL TRIAL: NCT00931411
Title: Double-Blind Study of Tolerance and Moisturizers Efficacy of Formulation 609580 20 Versus Formulation 609209 in Children With Atopic Dermatitis Under Normal Conditions of Use
Brief Title: Tolerance and Efficacy of Formulation 609580 20 Versus Formulation 609209 in Children With Atopic Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients would improve naturally due to weather conditions
Sponsor: Cosmetique Active International (Industry)
Collaborators: Innovaderm Research Inc. (Other)
Responsible Party: Principal Investigator, Robert BISSONNETTE, President and Dermatologist, Cosmetique Active International
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LRP07019; CCER 08-09-009 (Other: Comité centrale d'éthique de la recherche)
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Results first posted 2011-02-03 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Vitamin B3
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation 609580 20 then 609209 (Experimental): Formulation 609580 20 cream is applied topically to the entire body twice a day, morning and evening, after bathing for 42 days. This is followed by the same application of formulation 609209 for 2 weeks. Dosage is at the discretion of the parent applying the cream to the child.
  Interventions: Other: Formulation 609580 20; Other: Formulation 609209 (Lipikar Baume)
- Formulation 609209 then 609580 20 (Active Comparator): Formulation 609209 cream is applied topically to entire body, twice a day, morning and evening, after bathing for 42 days. This is followed by the same application of formulation 609580 20 for 2 weeks. Dosage is at the discretion of the parent applying the cream to the child.
  Interventions: Other: Formulation 609580 20; Other: Formulation 609209 (Lipikar Baume)

INTERVENTIONS:
Other: Formulation 609580 20 — Moisturizer, applied topically to whole body, twice a day, morning and evening, after bathing.
Other: Formulation 609209 (Lipikar Baume) — Moisturizer, applied topically to whole body, twice a day, morning and evening, after bathing.
  Other Names: Lipikar Baume

SUMMARY:
Atopic dermatitis is one of the most frequent skin diseases. The disease is often worst during winter months when the skin is drier. Mild to moderate cases of atopic dermatitis are often controlled by a moisturizer alone. The use of moisturizers has been shown to have beneficial effects on atopic dermatitis. It can break the dry skin cycle by hydrating the upper layer of the skin which may prevent the recurrence of the disease and can reduce the use of cream or ointment medications such as corticosteroids. Formulation 609580 20 was developed to keep the moisturizing efficacy of formulation 609209 but to improve its tolerance and cosmetic acceptability (easier to apply, nicer texture, etc.). The new formulation contains the same quantity of shea butter and glycerin but in a different excipient (inactive substance) than the commercial product. In addition, vitamin B3 was added to see if it could help in reducing itching.

The purpose of this study is to determine the safety and efficacy of two study products in children with atopic dermatitis. One of the study products (formulation 609580 20) is not commercially available (outside of clinical trials such as this one). The other study product (formulation 609209) has been approved in Canada and is currently available commercially under the trade name Lipikar Baume.

For this study the child will be randomly assigned to one of the following two groups:

* Group 1: 50 children will receive formulation 609209, the commercial formula for 42 days and will receive formulation 609580 20, the new formula, for 14 days.
* Group 2: 50 children will receive formulation 609580 20, the new formula, for 42 days and will receive formulation 609209, the commercial formula, for 14 days.

DETAILED DESCRIPTION:
A randomized clinical trial performed at five (5) centers (Montreal, Laval, Quebec City, (Quebec); Markham, London (Ontario), Canada). One hundred (100) patients are enrolled in the study. Subjects and parent(s) or guardian are asked to present to the clinic for five (5) visits (Screening, D0, D7, D42, D56). Formulation 609580 20 or 609209 is applied twice a day (morning and evening) to the whole body for a total of 42 days and then there is a crossover between the two formulations.

Efficacy is evaluated at D0, D7 and D42 measured by SCORAD (scoring atopic dermatitis). Tolerance is evaluated by the investigator at D7, D42 and D56. Global efficacy is measured by parents and investigator at D7 and D42. Medical photographs (optional) of lesions are taken with patients consent at D0 and D42. A crossover between the two products occurs at day 42 so that cosmetic acceptability can be compared at D42 and D56. Skin examinations are performed at all visits. A quality of life questionnaire is filled out by the parent(s) at D0 and D42.

ELIGIBILITY:
Inclusion Criteria:

* 3-12 years of age
* Suffering from a mild to moderate atopic dermatitis that is amenable to treatment with moisturizer only
* SCORAD (scoring atopic dermatitis) of 10-30 at screening and Day 0
* Diagnosis of atopic dermatitis must meet Hanifin's criteria (at least 3 basic features and at least 3 minor features; please refer to appendix D)
* Atopic dermatitis has been, in the opinion of the investigator, stable for the past 28 days
* Subject with parents able to apply the study product twice a day (each morning and evening) for a 56 days period
* Subject with parents agreeing not to change their child's lifestyle during the study period (including their usual body hygiene product (soap), the number of baths and showers per day, the laundry detergent and fabric softener used to wash the child's clothes)
* Subject with parents agreeing that their child uses only the test product as body emollient on the whole body during the study period
* Subject with parents available to completely follow the study with their child
* Subject with parents able and willing to sign the informed consent form and to comply with the study regulations of this protocol

Exclusion Criteria:

* Subject has another dermatological condition that could interfere with clinical evaluation including infected atopic dermatitis lesions
* Subject has a previous history of allergy to cosmetic products or any ingredients of the tested formulations
* Subject has received any systemic treatment, including PUVA (psoralen ultraviolet A) therapy for atopic dermatitis within 28 days prior to screening
* Subject has received any topical immunomodulators for atopic dermatitis (such as pimecrolimus or tacrolimus) within 14 days of Day 0
* Subject has received phototherapy within 14 days of Day 0
* Subject intends to expose him/herself to the sun during the trial
* Subject has known allergy to any component of tested products
* Subject has used any experimental treatment within 14 days of Day 0
* Subject has used any topical corticosteroid of class I-IV within 14 days of Day 0

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research
Locations (5):
- Canada (5):
  - The Guenther Dermatology Research Center, London, Ontario
  - Lynderm Research, Markham, Ontario
  - Innovaderm Research Inc, Laval, Quebec
  - Innovaderm Research Inc, Montreal, Quebec
  - Centre de recherche dermatologique du Québec Métropolitain, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Period: First Intervention - 42 Days
Arm/Group | Formulation 609580 20 Then 609209 | Formulation 609209 Then 609580 20
Started | 35 | 38
Completed | 31 | 35
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Period: After Crossover - 14 Days (up to Day 56)
Arm/Group | Formulation 609580 20 Then 609209 | Formulation 609209 Then 609580 20
Started | 31 | 35
Completed | 31 | 34
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Formulation 609580 20 Then 609209 | Formulation 609209 Then 609580 20 | Total
Number analyzed (Participants) | 35 | 38 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 38 | 73
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.11 (2.83) | 6.66 (2.36) | 6.88 (2.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 27 | 46
  Male | 16 | 11 | 27
Region of Enrollment [Number; unit: participants]
  Canada | 35 | 38 | 73
SCORAD - Score Atopic Dermatitis [Mean (Standard Deviation); unit: Units on a scale] — SCORAD - Score Atopic Dermatis measures intensity of erythema/darkening, edema/papulation, oosing/crust, excoriation, lichenfinication/prurigo and dryness on a scale from 0-3 for a total of 18 points. This score is multiplided by 3.5 and added to 1/5 of the affected percent body surface area. The final score is added to the score from a 10-point pruritus visual analog scale (VAS) and a 10-point loss of sleep VAS. Best score is 0, worst score is 103.
  Example:
  * 18 * 3.5 = 63
  * 63 + 20 = 83
  * 83 + 10 + 10 = 103
  Units on a scale | 21.5 (4.8) | 21.2 (5.2) | 21.3 (5.0)
Quality of Life Questionnaire [Mean (Standard Deviation); unit: Units on a scale] — The effect of formulation 609580 20 to improve quality of life compared to formulation 609209 as measured by changes in the quality of life questionnaire score from Day 0 to Day 42. Scale from -46 (worse) to 46 (better).
  Units on a scale | 4.75 (10.2) | 9.25 (12.2) | 7.1 (11.4)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in SCORAD (Scoring Atopic Dermatitis) From Day 0
Description: The efficacy of formulation 609580 20 to provide relief to children with atopic dermatitis compared to formulation 609209 as measured by the changes in SCORAD at Day 7 and Day 42. It measures intensity of erythema/darkening, edema/papulation, oozing/crust, excoriation, lichenfinication/prurigo and dryness on a scale from 0-3 for a total of 18 points. This score is multiplided by 3.5 and added to 1/5 of the affected percent body surface area. The final score is added to the score from a 10-point pruritus visual analog scale (VAS) and a 10-point loss of sleep VAS. Best score is 0, worst is 103.
Time Frame: 7 , 42 days
Population: All subjects that had at least one evaluation after the Day 0 visit were included in the efficacy evaluations if their overall compliance was between 70 and 120%. Missing data were replaced using the last observation carried forward (LOCF) method. Two patients lost to follow-up and 5 less than 70% compliant were not included in this analysis.
Measure: Mean (Standard Deviation); unit: Percentage of change in SCORAD
Groups:
- Formulation 609580 20: Formulation 609580 20 cream is applied topically to the entire body twice a day, morning and evening, after bathing for 42 days. Dosage is at the discretion of the parent applying the cream to the child.
- Formulation 609209: Formulation 609209 cream is applied topically to entire body, twice a day, morning and evening, after bathing for 42 days. Dosage is at the discretion of the parent applying the cream to the child.
Arm/Group | Formulation 609580 20 | Formulation 609209
Number analyzed (Participants) | 31 | 35
Percentage of change in SCORAD
  Day 7 | -35.5 (23.30) | -49.72 (24.62)
  Day 42 | -56.56 (36.92) | -61.99 (34.22)

2. Secondary Outcome: Change in Mean Global Efficacy (by Investigator).
Description: The efficacy of formulation 609580 20 to provide relief to children with atopic dermatitis compared to formulation 609209 as measured by the global efficacy evaluation scale at Day 7 and Day 42 (by investigator).
  * 0 = worsening
  * 1 = No change
  * 2 = Mild Improvement
  * 3 = Moderate Improvement
  * 4 = Good Improvement
  * 5 = Excellent Improvement
Time Frame: 7, 42 Days
Population: All subjects with all evaluations after the Day 0 visit were included in this evaluation if their overall compliance was >70 and <120%. Missing data were imputed using last observation carried forward (LOCF). Two patients lost to follow-up, one missing Day 7 value and 5 less than 70% compliant were not included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Formulation 609580 20 | Formulation 609209
Number analyzed (Participants) | 30 | 35
Units on a scale
  Day 7 | 3.23 (1.22) | 3.48 (1.22)
  Day 42 | 3.87 (1.5) | 4.06 (1.3)

3. Secondary Outcome: Change in Mean Global Efficacy (by Parent)
Description: The efficacy of formulation 609580 20 to provide relief to children with atopic dermatitis compared to formulation 609209 as measured by the global efficacy evaluation scale at Day 7 and Day 42 (by parent).
  * 0 = worsening
  * 1 = No change
  * 2 = Mild Improvement
  * 3 = Moderate Improvement
  * 4 = Good Improvement
  * 5 = Excellent Improvement
Time Frame: 7, 42 days
Population: All subjects with all evaluations after the Day 0 visit were included in this evaluation if their overall compliance was >70 and <120%. Missing data were imputed using last observation carried forward (LOCF). Two patients lost to follow-up, two missing Day 7 value and 5 less than 70% compliant were not included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Formulation 609580 20 | Formulation 609209
Number analyzed (Participants) | 30 | 34
Units on a scale
  Day 7 | 3.27 (1.14) | 3.06 (1.28)
  Day 42 | 3.8 (1.4) | 3.68 (1.3)

4. Secondary Outcome: Change in Mean Quality of Life
Description: The effect of formulation 609580 20 to improve quality of life compared to formulation 609209 as measured by changes in the quality of life questionnaire score from Day 0 to Day 42. Scale from -46 (worst) to 46 (best).
Time Frame: 0, 42 days
Population: All subjects with at least one evaluation after the Day 0 visit were included in this evaluation if their overall compliance between 70 and 120%. Missing data were imputed using last observation carried forward (LOCF). Two patients lost to follow-up, and 5 less than 70% compliant were not included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Formulation 609580 20 | Formulation 609209
Number analyzed (Participants) | 31 | 35
Units on a scale | 23.74 (12.74) | 23.09 (12.62)

5. Secondary Outcome: Change in Mean Cosmetic Acceptability Before Crossover
Description: The cosmetic acceptability of formulation 609580 20 compared to formulation 609209 as measured by the total score in the cosmetic acceptability questionnaire during the first 42 prior to the crossover. Scale from 44 (worst) to -44 (best).
Time Frame: 0, 42 days
Population: All subjects with at least one evaluation after the Day 0 visit were included in the cosmetic evaluation if their overall compliance between 70 and 120%. Missing data were imputed using last observation carried forward (LOCF). Two patients lost to follow-up, and 5 less than 70% compliant were not included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Formulation 609580 20 | Formulation 609209
Number analyzed (Participants) | 31 | 35
Units on a scale | -19.4 (10.4) | -20.4 (10.4)

6. Secondary Outcome: Change in Mean Cosmetic Acceptability After Crossover
Description: The cosmetic acceptability of formulation 609580 20 compared to formulation 609209 as measured by the total score in the cosmetic acceptability questionnaire during the 2 week period after the crossover. Scale from 44 (worst) to -44 (best). The 14 Days after the crossover is the same as Day 56 in the study.
Time Frame: 14 days (Day 42 to Day 56 of the study)
Population: Subjects that had at least one evaluation after the Day 0 visit were in analysis if they had overall compliance between 70 and 120%. Missing data were imputed using last observation carried forward. Two patients lost to follow-up, 1 early term and 5 less than 70% compliant were not included in this analysis and participants swapped after crossover.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Formulation 609580 20: Formulation 609580 20 cream is applied topically to the entire body twice a day, morning and evening, after bathing for 14 days after the crossover. Dosage is at the discretion of the parent applying the cream to the child.
- Formulation 609209: Formulation 609209 cream is applied topically to entire body, twice a day, morning and evening, after bathing for the 14 days after the crossover. Dosage is at the discretion of the parent applying the cream to the child.
Arm/Group | Formulation 609580 20 | Formulation 609209
Number analyzed (Participants) | 34 | 31
Units on a scale | -19.7 (13.3) | -17.8 (14.4)

7. Secondary Outcome: Change in Tolerance Before Crossover
Description: Tolerance of study products assessed by investigator at Day 7, 42. It was evaluated using the following scale:
  * 1) Very good tolerance: no objective or subjective intolerance during the study
  * 2) Good tolerance: very occasional symptoms, not resulting in cessation of applications, no objective sign
  * 3) Average tolerance: repeated symptoms of intolerance, no cessation of application and no objective sign
  * 4) Poor tolerance: symptoms requiring cessation of application, no objective sign
  * 5) Very poor tolerance: objective signs of irritative or allergic dermatitis
Time Frame: 7, 42 days
Population: All subjects that had at least one evaluation after the Day 7 (no Day 0 visit for this parameter) visit were included in the efficacy evaluations. Missing data were replaced using the last observation carried forward (LOCF) method. Four patients had no Day 7 visit to carry forward and were not included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Formulation 609580 20 | Formulation 609209
Number analyzed (Participants) | 34 | 35
Units on a scale
  Day 7 | 1.35 (0.60) | 1.60 (0.77)
  Day 42 | 1.38 (0.82) | 1.37 (0.81)

8. Secondary Outcome: Change in Mean Tolerance After Crossover
Description: Tolerance of study products assessed by investigator during the 2 weeks following the crossover (Day 56 of the study):
  * 1) Very good tolerance: no objective or subjective intolerance during the study
  * 2) Good tolerance: very occasional symptoms, not resulting in cessation of applications, no objective sign
  * 3) Average tolerance: repeated symptoms of intolerance, no cessation of application and no objective sign
  * 4) Poor tolerance: symptoms requiring cessation of application, no objective sign
  * 5) Very poor tolerance: objective signs of irritative or allergic dermatitis
Time Frame: 14 Days (Day 42 to Day 56 of the study)
Population: All subjects that had at least one evaluation after Day 7 (no day 0 visit for this parameter) were included in the analysis. Missing data were replaced using the last observation carried forward method. The same patients as in outcome #7 did not have results to carry forward and were not included in analysis (subjects swapped after crossover).
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Formulation 609580 20: Formulation 609580 20 cream is applied topically to the entire body twice a day, morning and evening, after bathing for the 14 days after the crossover. Dosage is at the discretion of the parent applying the cream to the child.
Arm/Group | Formulation 609580 20 | Formulation 609209
Number analyzed (Participants) | 35 | 34
Units on a scale | 1.66 (0.94) | 1.44 (0.66)

9. Secondary Outcome: Preferred Formulation
Description: Number of participants that preferred one formulation over the other. All patients started the study with one cream and crossed over to the other cream at Day 42 for another 14 days. Participants were asked which they prefered.
Time Frame: 56 days
Population: All subjects with an evaluation after the Day 42 visit were included in this evaluation if their overall compliance was between 70 and 120%. Two patients lost to follow-up, one with no Day 56 value and 5 less than 70% compliant were not included in this analysis.
Measure: Number; unit: Participants
Arm/Group | All Study Patients
Number analyzed (Participants) | 65
Participants
  Formulation 609580 20 | 35
  Formulation 605209 | 26
  No Preference | 4

ADVERSE EVENTS:
Time Frame: 56 days between the date of the first application and the final date of the study regardless of their compliance or their completion of the study.
Groups:
- Formulation 609580 20: Adverse events that were recorded before Day 42 for the group "Formulation 609580 20 then 609209" and recorded in the subsequent 2 weeks for the group "Formulation 609209 then 609580 20". Since this treatment was applied to both groups during this crossover study then the number of patients at risk for each treatment was the total of both groups.
- Formulation 609209: Adverse events that were recorded before Day 42 for the group "Formulation 609209 then 609580 20" and recorded in the subsequent 2 weeks for the group "Formulation 609580 20 then 609209". Since this treatment was applied to both groups during this crossover study then the number of patients at risk for each treatment was the total of both groups.
Arm/Group | Formulation 609580 20 | Formulation 609209
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/73
Other Adverse Events (participants affected / at risk) | 8/73 | 12/73
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Formulation 609580 20 (N=73) | Formulation 609209 (N=73)
Common cold (Infections and infestations) | 4 (4) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less